CLINICAL TRIAL: NCT01765296
Title: A Double-blind, Randomized, Multicenter, Active- and Placebo-Controlled Phase III Study to Evaluate the Efficacy and Safety of CG100649 in Osteoarthritis Patients
Brief Title: Phase III Study of CG100649 in Osteoarthritis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CG100649-3-01
Record Dates: First submitted 2013-01-08; First posted 2013-01-10 (Estimated); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Localized Primary Osteoarthritis of Hip; Localized Primary Osteoarthritis of Knee
Keywords: COX-1; COX-2; carbonic anhydrase; anti-inflammatory; Cyclooxygenase Inhibitors; Polmacoxib
MeSH Terms: interventions — CG100649; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Celecoxib (Active Comparator): Celecoxib 200 mg by mouth, once a day for 6 weeks (Treatment Phase), followed by CG100649 2 mg, oral, for 18 weeks (Safety Phase)
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator): Placebo capsule by mouth, once a day for 6 weeks (Treatment Phase), followed by CG100649 2 mg, oral, for 18 weeks (Safety Phase)
  Interventions: Drug: Placebo
- CG100649 (Experimental): CG100649 2 mg capsule by mouth, once a day for 6 weeks (Treatment Phase); CG100649 2 mg capsule by mouth, once a day for 18 weeks (Safety Phase)
  Interventions: Drug: CG100649

INTERVENTIONS:
Drug: CG100649 — 2 mg capsule
  Arms: CG100649
Drug: Celecoxib — 200 mg capsule
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Placebo — Mimic for CG100649 2 mg capsule and for celecoxib 200 mg capsule
  Arms: Placebo

SUMMARY:
* 6-week Efficacy Study The objective of this study is to prove the safety and non-inferiority of analgesic efficacy of CG100649 2 mg vs. celecoxib 200 mg, and analgesic superiority of CG100649 2 mg vs. placebo, when administered once a day in patients with osteoarthritis of the hip or knee over the 6 week Treatment period. The primary efficacy parameter is the difference from Baseline to Week 6 in the Western Ontario and McMaster Universities Index of Osteoarthritis (WOMAC)-Pain subscale.
* Extended Safety Study The objective of the Extended Safety Study is to collect a total of 24 weeks of safety data for CG100649 including the initial 6 weeks of safety data, and an additional 18 weeks of safety data for those subjects who agree on the consent form to continue into the Extended Safety Study. Subjects will be administered CG100649 2 mg only during 18 weeks of Extended Safety Study.

DETAILED DESCRIPTION:
1. Number of Subjects: 350 (2:2:1 ratio of experimental vs. active comparator vs. placebo comparator)
2. Adverse Events will be coded to preferred term and body system using the Medical Dictionary for Regulatory Activities (MedDRA)

ELIGIBILITY:
Inclusion Criteria (abbreviated)

1. Males or females, age 20 years or above, able and willing to provide written informed consent
2. Knee or Hip OA diagnosed according to American College of Rheumatology guidelines
3. Chronic pain for ≥3 months from OA
4. BP [systolic 90-140 mmHg, diastolic 50-90 mmHg] and pulse rate [resting 40-100 bpm].
5. WOMAC-Pain score in the index joint must be between 4-8 on a 0-10 numerical rating scale
6. Blood chemistry must be within 2x normal range
7. Urinalysis must be within normal limits; minor deviations are acceptable
8. Subjects and their sexual partners must agree to use double barrier contraception during the study period and for 3 months afterward, or be at least one year post- menopause, or provide proof of surgical sterility
9. For prior non-steroidal inflammatory drug (NSAID) users only, the subject has a history of positive therapeutic benefit
10. Subject is willing to limit alcohol intake to 2 or less drinks per day during study and the follow-up period
11. Subjects must be able to read, understand and follow study related documents.

Exclusion Criteria (abbreviated)

1. Use of any analgesics except the study medication or acetaminophen at any time
2. Use of any medications for ongoing chronic symptoms, or psychiatric disorders that could significantly diminish the cognitive ability or cause behavioral changes that would prevent the subject from complying with study procedures.
3. Subject is legally incompetent, or has active psychosis, or significant emotional problems which are sufficient to interfere with the conduct of the study
4. Use of anticoagulants (aspirin, warfarin, heparin, etc.) within 2 weeks of V1
5. Previous history of hypersensitivity or allergy to NSAIDs, COX-2 inhibitors, carbonic anhydrase inhibitors, sulfa drugs, aspirin, or acetaminophen/paracetamol
6. Subjects requiring knee or hip arthroplasty within 2 months of screening or anticipating any need for a surgical procedure on the index joint during the study
7. Diagnosed or treated for active GI ulcer, GI bleeding, ulcerative colitis, or severe renal, hepatic, or coagulant disorder within 6 months prior to randomization
8. History of nasal polyps, bronchospasm, urticaria, or anaphylactic shock
9. Subjects who have had surgery on the affected joint within 6 months prior to the study and subjects with a prosthesis at the index joint
10. Pregnant or breast-feeding, or expecting to conceive within the projected duration of the study
11. Subjects who are currently participating or have participated in other clinical studies within 4 weeks of screening or in any other clinical trial evaluating NSAIDs or COX-2 inhibitors within 6 months of screening
12. Subjects who have received even one dose of rofecoxib or etoricoxib at any time in their life
13. History of congestive heart failure with a status of New York Heart Association II-IV, ischemic heart disease, uncontrolled hypertension, peripheral arterial disease, cerebrovascular disease or subjects who have one of these diseases
14. Current user of recreational or illicit drugs or has had a recent history (1 year) of drug or alcohol abuse or dependence
15. History of neoplastic disease or chemotherapy within 5 years of V1, with the exception of non-metastatic skin cancer that has been completely cured
16. Subjects with gout, pseudogout, inflammatory arthritis, Paget's disease of bone, chronic pain syndrome, fibromyalgia, or another major joint disease
17. Subjects using i.v, i.m., or oral corticosteroids, i.a. steroids or hyaluronic acid injections within 1 month of V1
18. Subjects receiving a Chinese traditional arthritis treatment within 1 week of V1
19. Subjects who are not suitable to participate in the study by the investigator's clinical decision

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangsook Cho, Ph.D., Study Director — CrystalGenomics, Inc.
Locations (14):
- South Korea (14):
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - NHIC Ilsan Hospital, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Asan Medical Center, Seoul
  - Boramae Medical Center, Seoul
  - Ewha Womans University Hospital, Seoul
  - Inje University Seoul Paik Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
This medication already got NDA approval in Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | CG100649 | Celecoxib
Started | 71 | 146 | 145
Completed | 66 | 126 | 132
Not Completed | 5 | 20 | 13
Not completed — Protocol Violation | 0 | 5 | 4
Not completed — Withdrawal by Subject | 4 | 2 | 2
Not completed — Adverse Event | 1 | 13 | 5
Not completed — Lack of Efficacy | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | CG100649 | Celecoxib | Total
Number analyzed (Participants) | 71 | 146 | 145 | 362
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (8.97) | 62.5 (7.52) | 62.1 (7.59) | 62.4 (7.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 125 | 123 | 309
  Male | 10 | 21 | 22 | 53

OUTCOME MEASURES:

1. Primary Outcome: Change in WOMAC-Pain Subscale
Description: Western Ontario and McMaster Universities (WOMAC) OA index. Version 3.1 of the WOMAC knee and hip osteoarthritis index translated in Korean language will be used for each site enrolled in the trial.
  The numerical rating scale version of the WOMAC-Pain subscale was used, i.e., with the subject assessing each question by a 11-point (0-10) numerical rating scale, and the total pain score being represented by the sum of the 5 component item scores. A higher WOMAC score represented worse symptom severity, with 50 being the worst possible total score.
Time Frame: Baseline, Week 6
Population: Intent-to-Treat (ITT) population (Baseline Observation Carried Forward (BOCF))
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo administered orally, once a day for 6 weeks (Treatment Phase); During the extension, all participants received open-label CG100649 2 mg
- CG100649 2 mg: CG100649 2 mg capsule administered orally, once a day for 6 weeks (Treatment Phase); for 18 weeks (Safety Phase)
- Celecoxib 200 mg: Celecoxib 200 mg administered orally, once a day for 6 weeks (Treatment Phase); During the extension, all participants received open-label CG100649 2 mg
Arm/Group | Placebo | CG100649 2 mg | Celecoxib 200 mg
Number analyzed (Participants) | 71 | 146 | 145
units on a scale
  Baseline | 26.8 (4.58) | 27.9 (5.01) | 27.7 (5.08)
  Week 6 | 24.2 (7.41) | 22.7 (8.71) | 21.9 (7.65)
  Change From Baseline | -2.5 (6.73) | -5.3 (7.11) | -5.8 (6.67)
Statistical Analysis 1: Comparison: Placebo vs CG100649 2 mg; The primary efficacy outcome measure is the change in the WOMAC-Pain Subscale in the index joint at Week 6 vs. pre-dose Baseline and was analyzed using a mixed effect ANCOVA. Statistical tests to determine superiority between two treatment arms, CG100649 2 mg and placebo, are two-sided, and Non-inferiority between two treatment arms, CG100649 2 mg and celecoxib 200 mg is based on a one-sided 97.5% confidence interval of the difference; Test type: Non-Inferiority or Equivalence — The SD for the primary efficacy outcome measure (WOMAC-Pain Subscale in the index joint) has been assumed to be 11 units. A 10% between-group difference was chosen as the non-inferiority margin for this study. The following parameters were used to calculate the sample size needed for this non-inferiority study. * Level of significance, α = 0.025(one-sided) * Statistical power, 1-β = 0.95 * Difference between test group and comparison group, Δ=0, δ (>0) = non-inferiority margin; p = 0.011, ANCOVA
Statistical Analysis 2: Comparison: CG100649 2 mg vs Celecoxib 200 mg; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.425, ANCOVA

2. Secondary Outcome: Change of the WOMAC-physical Function Subscale at Week 3 and 6 From Pre-dose Baseline
Description: Western Ontario and McMaster Universities (WOMAC) OA index. Version 3.1 of the WOMAC knee and hip osteoarthritis index translated in Korean language will be used for each site enrolled in the trial.
  The 24 questions, which measure with 0-10 point numerical rating scale (NRS) with a maximum of 240 points to evaluate "Pain (5 questions)," "Stiffness (2 questions)," and "Physical Function (17 questions)" in WOMAC 3.1.
  Total scores for WOMAC-physical function is from 0 to 170 points. A higher WOMAC score represented worse symptom severity.
Time Frame: Baseline, Week 3 and Week 6
Population: Intent-to-Treat (ITT) (BOCF)
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | CG100649 2 mg | Celecoxib 200 mg
Number analyzed (Participants) | 71 | 146 | 145
units on a scale
  Week 3 | -5.7 [-10.6 to -0.8] | -13.7 [-17.5 to -9.9] | -10.7 [-14.5 to -6.9]
  Week 6 | -7.9 [-13.4 to -2.3] | -14.3 [-18.6 to -10.0] | -14.9 [-19.1 to -10.6]

ADVERSE EVENTS:
Time Frame: From ICF to Treatment Completion, up to 6 months (24weeks)
Groups:
- CG100649: CG100649 2 mg capsule administered orally, once a day for 6 weeks (Treatment Phase); for 18 weeks (Safety Phase)
- Celecoxib: Celecoxib 200 mg administered orally, once a day for 6 weeks (Treatment Phase); During the extension, all participants received open-label CG100649 2 mg
Arm/Group | Placebo | CG100649 | Celecoxib
Serious Adverse Events (participants affected / at risk) | 1/71 | 2/146 | 1/145
Other Adverse Events (participants affected / at risk) | 6/71 | 20/146 | 15/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=71) | CG100649 (N=146) | Celecoxib (N=145)
Colon adenoma (Villotubular adenoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=71) | CG100649 (N=146) | Celecoxib (N=145)
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 7 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 1 | 4
Oedema Peripheral (General disorders) | 0 | 7 | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) cannot provide any trial related information to external parties' without mutual agreement with the Sponsor. This is valid even after the contract is canceled.